CLINICAL TRIAL: NCT06474351
Title: Development and Fine-tuning of a Medical-grade Wearable Device with Interpretable Artificial Intelligence System for the Obstructive Sleep Apnea-hypopnea Syndrome (OSAHS) Screening
Brief Title: Developement of TipTraQ Home Sleep Test
Status: Completed | Type: Observational
Sponsor: PranaQ Pte. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: TipTraQ developement VGH
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The clinical study aims to develop and fine-tune the TipTraQ system, created by PranaQ, for home sleep apnea screening. The system comprises a wearable device and a cloud-based AI for estimating Total Sleep Time (TST) and Apnea-Hypopnea Index (AHI). This open-label, non-randomized study will recruit 240 subjects aged 20 and older from the Veteran General Hospital, Taipei.

DETAILED DESCRIPTION:
Sleep Breathing Disorders (SBD) is a common disorder in the population. However, a lot of patients are not aware of this disease and do not receive proper treatment, which not only impacts their personal health but also causes public disasters. Thus, a screening tool to find those patients becomes a critical point-of-care issue. To achieve this goal, a wearable device that is suitable for the screening is needed. The goal of this study is developing and fine-tuning a new sleep screening platform, TipTraQ, developed by PranaQ. TipTraQ is composed of a wearable device designed as a convenient screening device based on the photoplethysmography (PPG) technique and an interpretable artificial intelligent (AI) system that takes the PPG signal recorded by the wearable device as input and outputs and outputs estimated total sleep time (TST) and apnea-hypopnea index (AHI).

The study is open-label and non-randomized, planning to recruit 240 subjects. Participants will use the TipTraQ device alongside a companion mobile app, with data analysis supported by AI technology hosted on a cloud server. The TipTraQ device will be worn over fingertip. The primary goal is to assess the robustness of the TipTraQ system and fine-tuned the algorithm by comparing its output against the gold standard PSG annotations made by sleep experts.

ELIGIBILITY:
Inclusion Criteria:

Subjects from the age of 20 and older that have an indication for an in-lab PSG study. The subject should be able to understand the study and sign the informed consent before being enrolled in the study. During the study period, the subject can withdraw from the study any time.

Exclusion Criteria:

Subjects with the following medical conditions will be excluded from this study:

1. Heart transplant
2. Heart failure, New Youk Heart Association (NYHA) classification III or IV
3. Chronic opioid medication user Devastating Severe strokes, with the modified Rankin score (mRS)≥4
4. Tracheostomy
5. Incapable of comprehending and signing the informed consent and questionnaires, including but not limited to subjects with severe Alzheimer's, unconscious by head trauma, or of someone with limited mental capacity
6. Cannot correctly follow the order to use the TipTraQ device

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health or people who has indication to conduct polysomnography (PSG).
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index(AHI) | From the start of a single polysomnography study to the end of the recording. Usually range from 4 to 10 hours
  the combined average number of apneas and hypopneas that occur per hour of sleep
Oxygen Desaturation Index(ODI) | From the start of a single polysomnography study to the end of the recording. Usually range from 4 to 10 hours
  Average desaturation episodes with a decrease in the oxygen saturation of ≥4% or 3% per hour
Total Sleep Time(TST) | From the start of a single polysomnography study to the end of the recording. Usually range from 4 to 10 hours
  Total sleep time during the polysomnography (PSG)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taipei, Taiwan

REFERENCES:
- [Derived] Chen KW, Tseng CH, Lee HC, Liu WT, Chou KT, Wu HT. Validation of a fingertip home sleep apnea testing system using deep learning AI and a temporal event localization analysis. Sleep. 2025 May 12;48(5):zsae317. doi: 10.1093/sleep/zsae317. PMID 39821673